CLINICAL TRIAL: NCT03103776
Title: Involvement of Polyomaviruses in the Pathogenesis of Autoimmune Thyroiditis and Goitrigenesis.
Acronym: IPoTAIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0033
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Polyoma Virus Infection; Thyroiditis, Autoimmune
MeSH Terms: conditions — Polyomavirus Infections; Thyroiditis, Autoimmune | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who have Graves disease (Other)
  Interventions: Other: Comparison of Positive PCR Frequencies for Polyomavirus in Blood, Urine and / or Thyroid Tissue vs Basedow / Hashimoto
- Patients having a goiter (Other)
  Interventions: Other: Comparison of Positive PCR Frequencies for Polyomavirus in Blood, Urine and / or Thyroid Tissue vs Basedow / Hashimoto

INTERVENTIONS:
Other: Comparison of Positive PCR Frequencies for Polyomavirus in Blood, Urine and / or Thyroid Tissue vs Basedow / Hashimoto — Comparison of Positive PCR Frequencies for Polyomavirus in Blood, Urine and / or Thyroid Tissue vs Basedow / Hashimoto

SUMMARY:
Autoimmune thyroiditis and goitres are frequent pathologies.

DETAILED DESCRIPTION:
Autoimmune thyroiditis and goitres are frequent pathologies. On a predisposing genetic ground, environmental factors are potentially at their origin. Viral infections are the main factors involved in autoimmunity (herpes virus, viral hepatitis C, Erythrovirus B19 ..). However some viruses have an oncogenic potential and could be involved in goitrigenesis. It is also possible that some viruses are specifically implicated in the pathogenesis of Graves' disease or Hashimoto thyroiditis which combines goitre and autoimmunity.

The intrathyroidism of the viral genome of a polyomavirus, the BK virus, has recently been reported in patients with goitre or cancer. The BK virus is a small ubiquitous virus of 40 nm diameter with double-stranded DNA contained in a non-enveloped icosahedral capsid. It is mainly known for triggering renal and bladder pathologies including urothelial tumors in the immunocompromised patient, tubulo-interstitial nephropathy in the renal transplant patient, as well as hemorrhagic cystitis in the patient grafted to the bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient Age ≥ 18 years
* Patients referred to the ENT service of the CHU of Amiens for thyroidectomy in the context of a goitre, a Graves' disease or a thyroiditis of Hashimoto.
* Patients must have signed informed consent.
* Affiliation to a social security scheme

Exclusion Criteria:

* Minor Patients,
* Patient under tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Investigate the presence of BK Polyomavirus and compare the prevalence in patients operated with goitre or Grave or Hashimoto's disease | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France